CLINICAL TRIAL: NCT05194969
Title: Comparison of Wet-to-dry vs Petrolatum and Non-stick Dressing for Second Intention Healing Following Hidradenitis Suppurativa Surgery
Brief Title: Wet-to-dry vs Petrolatum & Non-stick Dressings After Hidradenitis Suppurativa Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 21-1989
Record Dates: First submitted 2022-01-05; First posted 2022-01-18 (Actual); Results first posted 2024-08-28 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2024-01

CONDITIONS: Hidradenitis Suppurativa; Surgical Wound
MeSH Terms: conditions — Hidradenitis Suppurativa; Surgical Wound

STUDY DESIGN:
Intervention Model Description: This study will be a randomized, blinded trial of two postoperative bandaging techniques: wet-to-dry dressings vs. petrolatum with non-stick bandaging.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Following the surgical procedure, the principal investigator (PI) will exit the exam room. The PI will not be present for bandaging administration and training and thus be blinded to the wound dressing technique. The patient will not be blinded as bandaging will be administered at home.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Wet-to-dry Dressings (Active Comparator): Participants in this arm will receive standard of care wet-to-dry dressings.
  Interventions: Device: Wet-to-Dry Dressings
- Petrolatum with Non-Stick Gauze (Experimental): Participants in this arm will receive petrolatum with non-stick gauze.
  Interventions: Device: Petrolatum with Non-Stick Gauze

INTERVENTIONS:
Device: Wet-to-Dry Dressings — This dressing technique involves moistening a piece of gauze with normal saline or other cleansing solution, placing the moistened gauze on the wound, allowing the gauze to dry, and then removing and replacing the bandage regularly over a period of days to weeks
  Arms: Wet-to-dry Dressings
Device: Petrolatum with Non-Stick Gauze — This dressing approach involves applying a thick layer of petrolatum to the wound once or twice daily to maintain a moist wound base. After placement of petrolatum, the wound is covered with nonadherent gauze and tape or another bordered dressing.
  Arms: Petrolatum with Non-Stick Gauze

SUMMARY:
Hidradenitis suppurativa (HS) is a chronic, severe, inflammatory skin disease associated with pain, drainage, odor, and disability characterized by recurring abscesses, nodules, and tunneling sinuses in intertriginous locations such as the groin, buttocks, and axillae. HS has more negative impact on patients' quality of life than all other common dermatologic diseases and is common, affecting ~1% of the general population, with higher risk for females (3:1) and Black patients. The onset is often in adolescence. As HS has been under-studied historically, there is an unmet medical need to develop more effective treatment for this disease. While many patients are managed with medications and lifestyle modifications alone, a subset of HS patients benefit from surgical intervention. Proper wound care following HS surgery is paramount, as facilitating proper healing and minimizing infection can prevent post-operative complications, morbidity and the need for future procedures. While many physicians continue to use wet-to-dry dressings as the standard of care for HS patients post-operatively, it is likely that the drawbacks of this dressing technique outweigh the benefits. This study hopes to answer the question of whether or not wet-to-dry dressings should truly be standard of care or whether an alternate form of wound dressings, such as petrolatum with non-stick bandaging, is at least equitable if not superior in effect, and associated with fewer drawbacks such as associated pain and time dedicated to dressing changes. This study will be a randomized, single-blind trial of two postoperative bandaging techniques: wet-to-dry dressings vs. petrolatum with non-stick bandaging. Primary outcomes will be tracked using the photographic wound assessment tool (PWAT), pressure ulcer scale of healing (PUSH) tool, and Wound Quality of Life (QOL) Survey. There is potential for this study to apply to surgical interventions outside of HS, as the study addresses the bandaging technique (wet-to-dry) that is standard of care after many surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Male & females > or = 16 years of age
* Patient must have undergone a standard-of-care surgical procedure for HS with planned secondary intention healing of the wound.
* Must be able to provide adequate informed consent for themselves
* Patient must be capable of performing either of the recommended wound care regimens on their own or have someone available to consistently assist with wound care.

Exclusion Criteria:

* Patients with surgically closed wounds (sutures, staples)
* Patients with preference for specific types of bandaging protocols
* Patients that have not been able to tolerate either wet-to-dry or petrolatum and non-stick bandages in the past

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Sayed, MD, Study Director — University of North Carolina, Chapel Hill; Franklin R Blum, BS, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC School of Medicine Department of Dermatology, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator who proposes to use the data has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Background] van der Zee HH, Jemec GB. New insights into the diagnosis of hidradenitis suppurativa: Clinical presentations and phenotypes. J Am Acad Dermatol. 2015 Nov;73(5 Suppl 1):S23-6. doi: 10.1016/j.jaad.2015.07.047. PMID 26470610
- [Background] von der Werth JM, Williams HC. The natural history of hidradenitis suppurativa. J Eur Acad Dermatol Venereol. 2000 Sep;14(5):389-92. doi: 10.1046/j.1468-3083.2000.00087.x. PMID 11305381
- [Background] Ring HC, Theut Riis P, Miller IM, Saunte DM, Jemec GB. Self-reported pain management in hidradenitis suppurativa. Br J Dermatol. 2016 Apr;174(4):909-11. doi: 10.1111/bjd.14266. Epub 2016 Jan 6. No abstract available. PMID 26521975
- [Background] Ingram JR, Jenkins-Jones S, Knipe DW, Morgan CLI, Cannings-John R, Piguet V. Population-based Clinical Practice Research Datalink study using algorithm modelling to identify the true burden of hidradenitis suppurativa. Br J Dermatol. 2018 Apr;178(4):917-924. doi: 10.1111/bjd.16101. Epub 2018 Feb 22. PMID 29094346
- [Background] Augustin M, Conde Montero E, Zander N, Baade K, Herberger K, Debus ES, Diener H, Neubert T, Blome C. Validity and feasibility of the wound-QoL questionnaire on health-related quality of life in chronic wounds. Wound Repair Regen. 2017 Sep;25(5):852-857. doi: 10.1111/wrr.12583. Epub 2017 Nov 2. PMID 29080332
- [Background] Stotts NA, Rodeheaver GT, Thomas DR, Frantz RA, Bartolucci AA, Sussman C, Ferrell BA, Cuddigan J, Maklebust J. An instrument to measure healing in pressure ulcers: development and validation of the pressure ulcer scale for healing (PUSH). J Gerontol A Biol Sci Med Sci. 2001 Dec;56(12):M795-9. doi: 10.1093/gerona/56.12.m795. PMID 11723157
- [Background] Thompson N, Gordey L, Bowles H, Parslow N, Houghton P. Reliability and validity of the revised photographic wound assessment tool on digital images taken of various types of chronic wounds. Adv Skin Wound Care. 2013 Aug;26(8):360-73. doi: 10.1097/01.ASW.0000431329.50869.6f. PMID 23860221
- [Background] Eaglstein WH, Davis SC, Mehle AL, Mertz PM. Optimal use of an occlusive dressing to enhance healing. Effect of delayed application and early removal on wound healing. Arch Dermatol. 1988 Mar;124(3):392-5. PMID 3345089
- See also: PUSH Tool — https://cdn-links.lww.com/permalink/jwocn/a/jwocn_38_4_2011_04_07_gardner_1_sdc1.pdf
- See also: Wound QOL Survey — https://www.daemen.edu/sites/default/files/Wound-Outcome-Measure-Questionnaire.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Wet-to-dry Dressings | Petrolatum With Non-Stick Gauze
Started | 39 | 35
Completed | 27 | 26
Not Completed | 12 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Wet-to-dry Dressings | Petrolatum With Non-Stick Gauze | Total
Number analyzed (Participants) | 39 | 35 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (14.5) | 34.8 (9.5) | 37.8 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 26 | 57
  Male | 8 | 9 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 38 | 34 | 72
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 24 | 42
  White | 16 | 10 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 0 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39 | 35 | 74
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] | 37.6 [23.3 to 60.2] | 37.0 [21.9 to 64.3] | 37.3 [21.9 to 64.3]
Smoking History [Count of Participants; unit: Participants]
  Current Smoker | 5 | 2 | 7
  Former Smoker | 6 | 7 | 13
  Never Smoker | 28 | 26 | 54
Hurley Stage [Count of Participants; unit: Participants] — Hurley Stage 1: disease limited to inflammatory nodules and abscesses without significant scars or tunnels. Hurley Stage 2: inflammatory nodules, abscesses, and 1 or limited draining tunnels or scars. Hurley Stage 3: inflammatory nodules, abscesses, and multiple or extensive tunnels and/or scars
  Participants
    Hurley I | 0 | 0 | 0
    Hurley II | 26 | 22 | 48
    Hurley III | 13 | 12 | 25
    Hurley Unreported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Wound QOL Survey Score Over Time
Description: A validated Wound Quality of Life (QOL) Survey will be administered that focuses on patient-reported outcomes of level of wound pain, pain with dressing changes (application and removal), satisfaction with the bandaging, and ease of application of the bandaging, all 17 elements on a 0-4 scale. A mean score is calculated using each component such that a total score ranges from 0 to 4 with higher scores indicating a worse outcome.
Time Frame: Administered at 1, 2, 4 and 6 weeks post-surgery
Population: All available data are reported. Unreported data are for those lost to follow-up.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Wet-to-dry Dressings | Petrolatum With Non-Stick Gauze
Number analyzed (Participants) | 33 | 30
score on a scale
  Week 1 | 1.14 [0.1 to 3.1] | 0.94 [0.0 to 3.3]
  Week 2 | 0.77 [0.0 to 3.5] | 0.66 [0.0 to 2.6]
  Week 4: number analyzed (Participants) | 27 | 27
  Week 4 | 0.51 [0.0 to 1.9] | 0.54 [0.0 to 2.6]
  Week 6: number analyzed (Participants) | 24 | 26
  Week 6 | 0.28 [0.0 to 0.9] | 0.42 [0.0 to 2.9]

2. Primary Outcome: PUSH Score Over Time
Description: The pressure ulcer scale for healing (PUSH) tool is a validated means of measuring wound healing over time, specifically wounds that heal via secondary intent, by taking into account things like wound size and wound exudate, among others. Scores range from 0-17 with higher scores indicating inferior wound healing.
Time Frame: Completed at 1, 2, 4 and 6 weeks post-surgery utilizing images submitted by patients
Population: All available data are reported. Unreported data are for those lost to follow-up.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Wet-to-dry Dressings | Petrolatum With Non-Stick Gauze
Number analyzed (Participants) | 24 | 21
score on a scale
  Week 1 | 11.0 [5.0 to 15.0] | 11.4 [5.0 to 14.0]
  Week 2 | 9.1 [0.0 to 14.0] | 10.0 [4.0 to 14.0]
  Week 4 | 5.7 [0.0 to 13.0] | 6.2 [0.0 to 12.0]
  Week 6 | 3.9 [0.0 to 11.0] | 2.7 [0.0 to 8.0]

3. Primary Outcome: Pain With Dressing Changes Over Time
Description: The numeric rating scale (NRS) will be used, where patients will be asked to rate pain with dressing changes and general pain on a scale from 0-10 with higher scores indicating worse pain. This information will be collected in the patient survey that is sent post-operatively.
Time Frame: Collected at 1, 2, 4 and 6 weeks post-surgery
Population: All available data are reported. Unreported data are for those lost to follow-up.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Wet-to-dry Dressings | Petrolatum With Non-Stick Gauze
Number analyzed (Participants) | 33 | 30
score on a scale
  Week 1 Pain with Dressing Removal | 6.2 [0 to 10] | 3.6 [0 to 10]
  Week 2 Pain with Dressing Removal | 3.5 [0 to 10] | 2.3 [0 to 8]
  Week 4 Pain with Dressing Removal: number analyzed (Participants) | 27 | 27
  Week 4 Pain with Dressing Removal | 2.1 [0 to 10] | 1.6 [0 to 7]
  Week 6 Pain with Dressing Removal: number analyzed (Participants) | 25 | 26
  Week 6 Pain with Dressing Removal | 1.4 [0 to 10] | 1.1 [0 to 8]
  Week 1 Pain with Dressing Application | 3.0 [0 to 8] | 2.1 [0 to 7]
  Week 2 Pain with Dressing Application | 2.2 [0 to 7] | 1.3 [0 to 6]
  Week 4 Pain with Dressing Application: number analyzed (Participants) | 27 | 27
  Week 4 Pain with Dressing Application | 1.2 [0 to 7] | 1.0 [0 to 6]
  Week 6 Pain with Dressing Application: number analyzed (Participants) | 25 | 26
  Week 6 Pain with Dressing Application | 0.5 [0 to 7] | 0.7 [0 to 6]

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent through 6 weeks post-surgery.
Arm/Group | Wet-to-dry Dressings | Petrolatum With Non-Stick Gauze
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/35
Other Adverse Events (participants affected / at risk) | 1/39 | 0/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wet-to-dry Dressings (N=39) | Petrolatum With Non-Stick Gauze (N=35)
Prolonged bleeding during dressing changes (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-01): https://cdn.clinicaltrials.gov/large-docs/69/NCT05194969/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/69/NCT05194969/ICF_001.pdf